CLINICAL TRIAL: NCT06287567
Title: An Open-label, Single-arm Study to Evaluate the Efficacy and Safety of Lusutrombopag in Chinese Adults With Persistent or Chronic Immune Thrombocytopenia
Brief Title: Lusutrombopag in the Treatment of Immune Thrombocytopenia (ITP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023078
Record Dates: First submitted 2024-02-01; First posted 2024-03-01 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Idiopathic Thrombocytopenic Purpura; Immune Thrombocytopenia
Keywords: Lusutrombopag; Immune thrombocytopenia; Thrombopoietin receptor agonists
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — lusutrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Lusutrombopag (Experimental): Participants receive lusutrombopag 3 mg administered orally once a day for up to 4 weeks and titrated to a maximum dose of 6 mg during week 5 and week12 based on the platelet count (PLT)
  Interventions: Drug: Lusutrombopag Oral Tablet

INTERVENTIONS:
Drug: Lusutrombopag Oral Tablet — Participants receive lusutrombopag 3 mg administered orally once a day for up to 4 weeks and doses are adjusted based on platelet counts during week 5-12. If a subject's platelet count remains < 50x10^9 /L, the dose could have been increased up to a maximum dose of 6 mg（2 tablets).If a subject's platelet count reaches ≥ 250x10^9 /L during the first 4 weeks, treatment is stopped and participants are allowed to enter into Titration Study in advance when platelet count drops to ≥100x10^9 /L.
  Other Names: MULPLETA®; S-888711

SUMMARY:
This exploratory study is to investigate the efficacy, safety and tolerability of Lusutrombopag in the treatment of primary immune thrombocytopenia in Chinese patients who have failed first-line therapy

DETAILED DESCRIPTION:
This is an open-label, single-arm study of lusutrombopag initiated at a dose of 3mg daily titrated to a maximum dose of 6mg daily in the treatment of Chinese adults with persistent or chronic Immune thrombocytopenia (ITP) with or without prior splenectomy after failing first line therapy such corticosteroids and IV immunoglobulin. The study consists of three phases: Screening, Core Study（participants are treated with lusutrombopag 3mg daily for up to 4 weeks), and Titration study (participants are treated with lusutrombopag titrated to a maximum dose of 6mg daily according to their platelet counts）

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥18 years of age
2. Subjects>60 years must have had a diagnostic bone marrow aspiration in the last 3 years or responded to treatment (platelet count ≥50 x 10^9/L)
3. Participants diagnosed with primary persistent/chronic ITP (greater than or equal to 3 months duration) and an average of two platelet count less than 30 x 10^9/L. Conditions which may cause thrombocytopenia other than ITP should be ruled out, including but not limited to systemic lupus erythematosus (SLE)，aplastic anemia (AA), and myelodysplastic syndromes (MDS)
4. Relapsed persistent or chronic ITP status, with or without prior splenectomy. Participants who previously received one or more ITP therapies
5. Subjects receiving rescue therapy (including but not limited to corticosteroids, immunoglobulins and immunosuppressant) must have completed these therapies for at least 1 week or failed within 1 week prior to dosing on the first day (Visit 1)
6. Subjects receiving stable dosages of cyclosporine A, mycophenolate mofetil, azathioprine, or danazol are allowed, but must be receiving a dose that has been stable for at least 4 weeks prior to dosing on the first day (Visit 1)
7. Subjects receiving Chinese herbal medicine must be stopped 1 weeks prior to dosing on the first day (Visit 1), and Chinese herbal medicine is not allowed during the study
8. Subjects receiving steroid therapy must be on a stable dose for at least 2 weeks prior to screening (same milligram amount ± 10%； and ≤20 mg of equivalent dose of prednisone)
9. Two consecutive mean platelet count < 30×10^9/(a single platelet count of< 35×10^9/L is allowed） during screening if subjects were not receiving steroids, or two consecutive mean platelet count < 50×10^9/ if they were receiving steroids. Two Platelet counts must be measured at an interval of greater than 2 days and less than 14 days，and the second platelet count must be measured within 96 hours of day1（Visit 1）
10. Prothrombin time (PT) and activated partial thromboplastin time (APTT) within 20% of the upper limit of normal (ULN) at Screening or PT did not exceed normal value by ±3s and APTT by ±10s. No other history of coagulation state except ITP.
11. A complete blood count within the reference range ，including count of white blood cell (WBC) differential not indicative of a disorder other than ITP, with the following exceptions: a) Hemoglobin: participants with hemoglobin levels between 10 g/dL (100 g/L) and the lower limit of normal (LLN) are eligible for inclusion; participants with anemia(hemoglobin levels <10g/dl ) clearly attributable to ITP (excessive blood loss) are also eligible for inclusion; b) Absolute neutrophil count (ANC) greater than or equal to 1.5x10^9/L (elevated WBC/ANC due to corticosteroid treatment is acceptable).
12. All subjects must agree to take progestin or barrier contraception: patients with potential fertility (excluding hysterectomy, bilateral salpingectomy, bilateral tubal ligation or postmenopausal women for more than one year; Men with bilateral vasectomy) must take effective contraceptive measures at least 2 weeks before taking the study drug for the first time, throughout the study and within 28 days after the end of the study (or early termination of the study); Women with potential fertility must have a negative pregnancy test during the screening period and on the 0th day of the trial.
13. A signed and dated written consent obtained prior to the performance of Screening procedures

Exclusion Criteria:

1. History of inherited or acquired, clinically important hemorrhagic clotting disorder
2. Females who were pregnant or lactating, or receiving other hormone/chemical contraceptives
3. Patients with potential fertility refused to take contraceptive methods
4. Laboratory abnormalities

   * Hemoglobin <10.0 g/dL for men or women, not clearly related to ITP
   * Absolute neutrophil count < 1000/mm3
   * Abnormal peripheral blood smear with evidence of fibrosis confirmed by bone marrow biopsy
   * Total bilirubin > 1.5 x ULN
   * Alanine aminotransferase (ALT) > 1.5 x ULN
   * Aspartate aminotransferase (AST) > 1.5 x ULN
   * Creatinine > 1.5 x ULN
   * Human immunodeficiency virus positive
   * Hepatitis A Immunoglobulin M（IgM) antibody positive, hepatitis B surface antigen positive and HBV DNA ≥1000IU/ml or hepatitis C antibody positive，with a history of acute hepatitis, cirrhosis, portal hypertension or chronic active hepatitis.
   * Thyroid stimulating hormone (TSH) > 1.5 x ULN; or
   * Free thyroxine (T4) > 1.5 x ULN
5. Exposure to previous thrombopoietin (TPO) mimetics/agonists (e.g. romiplostim, recombinant human thrombopoietin (rhTPO), avatrombopag, eltrombopag and herombopag) within 4 weeks prior to initial screening.In addition, participants are allowed to be enrolled at the discretion of the investigator when platelet counts are below 30 x 10^9/L within the 4 weeks after withdrawal of thrombopoietin (TPO) mimetics/agonists
6. Subjects unresponsive to previous TPO mimetics/agonists
7. Exposure to an investigative medication within 4 weeks prior to the initial Screening Visit or Use of the following drugs or treatment prior to Visit 1 (Day 1):

   * Within 12 weeks - alemtuzumab, multi-drug systemic chemotherapy, stem cell therapy
   * Within 12weeks - rituximab
8. History of clinically significant cardiovascular or thromboembolic disease within 26 weeks prior to Initial screening
9. Splenectomy within 4 weeks prior to Initial Screening
10. Other abnormalities except ITP or situations that investigators deem inappropriate to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with a Platelet Response after 4 Weeks | on Day 29 of Treatment
  Platelet responses to lusutrombopag was evaluated using the platelet count defined as ≥50x10^9 /L on study drug treatment after 4 weeks of dosing（on Day 29) or prematurely ≥250x10^9 /L prior to Day 29.

SECONDARY OUTCOMES:
Percentage of Participants with a Platelet Response after 12 Weeks (Day 85) | on Day 85 of treatment
  Platelet responses to lusutrombopag was evaluated using the platelet count defined as ≥50x10^9 /L on study drug treatment after 12 weeks of dosing（on Day 85).
Percentage of Participants Who Achieved a Platelet Count of ≥50×10^9/L After 6 Weeks of Dosing | on Day 43 of treatment
  Platelet responses to lusutrombopag was evaluated using the platelet count defined as ≥50x10^9 /L after week 6
Percentage of Participants Who at least once Achieved a Platelet Count of ≥50x10^9/L in Week 1 ,2,3,4 in the Core Study | Baseline, Week 4
  Platelet responses to lusutrombopag was evaluated using the platelet count defined as ≥50x10^9 /L from baseline to Week 4.
Change in Platelet Count | Baseline, 12 Weeks
  Change from baseline in platelet count was assessed at every visit from Baseline to Week 12
Percentage of Participants Who at least once Achieved a Platelet Count of≥50x10^9 /L during the Treatment | Baseline, up to 12 Weeks
  Platelet responses to lusutrombopag was evaluated using the platelet count defined as ≥50x10^9 /L. Participants who at least once achieved a platelet count of ≥50x10^9 /L during the Core Study and Titration Study respectively were assessed.
Percentage of Participants Who at least once Achieved a Platelet Count of≥100x10^9 /L during the treatment | Baseline, up to 12 Weeks
  Platelet's complete responses to lusutrombopag was evaluated using the platelet count defined as a platelet count ≥100x10^9 /L. Participants who at least once achieved a platelet count of ≥100x10^9 /L during the Core Study and Titration Study respectively were assessed.
Time to first Achieve a Platelet Count of ≥ 50x10^9/L | Baseline, up to 12 Weeks
  The time to first achieve a response was defined as the Day when participants first reached a platelet count of ≥ 50×10^9/L from baseline.
Time to first Achieve a Platelet Count of ≥100x10^9 /L | Baseline, up to 12 Weeks
  Defined as the Day when participants first reached a platelet count of ≥ 100×10^9/L from baseline.
Percentage of Participants Who at least once Achieved a Platelet Coun platelet count≥30×10^9/L, a≥2-fold increase from baseline within week 1-4 and week 5-12，respectively. | Baseline, up to 12 Weeks
  The percentage of partial response were defined as a platelet count of ≥30×10^9/L, a≥2-fold increase from baseline
Durable Platelet Response (platelet count ≥50×10^9/L in ≥75% of weeks) Rate | Baseline, up to 12 Weeks
  Durable platelet response rate was defined as platelet count ≥50×10^9/L in ≥75% of assessments(weeks)
Cumulated Number of Weeks of Response（≥50x10^9/L） | Baseline, up to 12 Weeks
  Cumulative number of weeks of platelet response was defined as the total number of weeks in which platelet count is ≥50x10^9/L during the Core Study and Titration Study
Percentage of Participants with a Reduction in the use of Concomitant ITP Medications from Baseline | Day 29，Week 12
  Lusutrombopag dose titration and downward titration of concomitant ITP medications was allowed at Week ,when Titration Study begins.
The Incidence and Rating of Bleeding Events During the Study | Baseline，Week12
  Bleeding assessments were performed by the Investigator according to the World Health Organization (WHO) criteria bleeding scale:
  Grade 0: no bleeding; Grade 1: petechial bleeding; Grade 2: mild blood loss (clinically significant); Grade 3: gross blood loss, requires transfusion (severe); Grade 4: debilitating blood loss, retinal or cerebral associated with fatality.
Percentage of Participants Who Required Rescue Therapy for Bleeding During the Study | Baseline , Week16
  Participants who received rescue therapy for bleeding events during the study. steroids, intravenous immunoglobulin and platelet transfusion were considered as rescue therapy for bleeding events.
Number of Participants With Adverse Events (AEs) | Baseline through Week 12 while receiving treatment and at Week 16 after discontinuation of treatment.
  An AE is defined as any untoward medical occurrence in a subject administered a pharmaceutical product during the course of a clinical investigation, including any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product (IP), whether or not thought to be related to the IP. AEs reported after initial study drug administration were considered treatment-emergent.
  A serious adverse event is defined as any AE that resulted in death, was life-threatening, hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, or a congenital anomaly/birth defect or an important medical event that, based upon medical judgment, may jeopardize the participant or require medical or surgical intervention to prevent one of the outcomes listed above.
  A treatment-related AE is any AE determined by the investigator to be possibly related, probably related, or definitely related to study drug.
Change in Health-related Quality of Life Assessed by FACIT-F Scale from Baseline to Week 16 | Baseline，Week16
  The Functional Assessment of Chronic Illness Therapy-Fatigue scale (FACIT-F) assesses the severity of patient's fatigue. The Full version of FACIT-F contains 40 items. Total score is computed by summing 5 subscales: ranging from 0-160.This study assessed the subscale Fatigue (range 0-52), which contains 13 items, The higher the score, the milder the patients' fatigue.
Change in Health-related Quality of Life Assessed by ITP-PAG Scale from Baseline to Week 16 | Baseline，Week16
  The Immune Thrombocytopenic Purpura (ITP)-Patient Assessment Questionnaire (ITP-PAG) assesses the overall quality of life (Qol) of patients. Possible scores range from 0 to 100. Higher total score indicates better QoL

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Lei, MD, Principal Investigator — Chinese Academy of Medical Science and Blood Disease Hospital
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China